CLINICAL TRIAL: NCT00008476
Title: Evaluation of Vanilloid Receptor Inactivation for Preemptive Analgesia
Brief Title: Capsaicin to Control Pain Following Third Molar Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 010056; 01-D-0056
Record Dates: First submitted 2001-01-09; First posted 2001-01-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-01

CONDITIONS: Facial Pain
Keywords: Preemptive Analgesia; Vanilloid; Vanilloid Receptor (VR); Capsaicin; Acute Pain; Orofacial; Visual Analog Scale (VAS); Resiniferatoxin; Healthy Volunteer; Wisdom Teeth; Pain
MeSH Terms: conditions — Facial Pain; Acute Pain; Pain | interventions — Capsaicin

INTERVENTIONS:
Drug: Capsaicin

SUMMARY:
This study will test the effectiveness of the drug capsaicin in controlling pain after third molar (wisdom tooth) extraction. Capsaicin, the ingredient in chili peppers that makes them "hot," belongs to a class of drugs called vanilloids, which have been found to temporarily inactivate pain-sensing nerves.

Healthy normal volunteers between 16 and 40 years of age who require third molar (wisdom tooth) extraction may be eligible for this study. Participants will undergo the following procedures in three visits:

Visit 1:

Patients will have touch (sensory) testing by the following three methods: 1) a warm sensor applied to the gums and the patient will rate when they first feel heat and when the heat feels painful; 2) the bristles of a small paint brush will be gently stroked across the gums, and the patient will say whether it feels painful; 3) a light touch will be applied to the gums with a small needle, and the patient will rate the pain intensity following the touch.

After testing, patients will be numbed with a local anesthetic (bupivacaine) and then capsaicin or placebo (an inactive solution) will be injected next to the tooth. The tooth then will be extracted one day later.

Visit 2:

Patients will return to the clinic after 24 hours to repeat the same type of sensory testing. After testing, patients will be sedated and numbed with a local anesthetic (lidocaine) and given an intravenous injection of either saline or ketorolac (30 mg). After the extraction, pain ratings will be recorded every 20 minutes, for up to 6 hours. During this time, patients will be monitored for numbness, pain, side effects and vital signs (heart rate, blood pressure, respiration, etc.). Those who request pain medicine will receive acetaminophen and codeine. Patients will be required to stay for up to 3 more hours after this and then they will then be discharged with pain medicine.

Visit 3:

Patients will return to the clinic after another 48 hours to repeat the same sensory testing. Remaining wisdom teeth will be removed "off-study" at least three weeks following the first visit.

DETAILED DESCRIPTION:
Successful preemptive analgesia strategies are superior to traditional pain management schemes in the management of post-operative pain. However, agents with appropriate pharmacokinetic properties are not readily available. The premise of this double-blind, placebo and positive-controlled clinical study is to evaluate the efficacy of vanilloid agonists as preemptive agents in an oral surgery tissue injury model. Vanilloids are a class of small organic compounds; the most familiar of which is capsaicin, the active ingredient in hot pepper. Binding of capsaicin to the vanilloid-1 receptor produces initial activation and then long-acting desensitization of pain specific neurons. We propose to produce a selective, long-term inactivation of peripheral pain transmission through the local application of capsaicin in the oral mucosa in an effort to prevent or reduce post-operative pain in the oral surgery model. Healthy subjects will be recruited, and following local anesthesia, will be given an intramucosal injection of either capsaicin or placebo. (Or as a positive control, 24 hours later, intravenous Toradol). Subjects will have one lower impacted wisdom tooth extracted under local anesthesia and then will rate their pain. The time of analgesic rescue medication request will be noted. A decrease in post-operative pain and decrease in analgesic use will be taken as a positive effect of the vanilloid for decreasing post-operative pain. We anticipate that through the long term blockade of pain specific fibers pre-operatively that there will be a significant attenuation of post-operative pain development following surgery. This has significant implications for reducing pain and suffering, decreasing analgesic use, and reducing post-operative complications following surgery.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female volunteers referred for mandibular third molar extraction with a minimal difficulty rating score of 3-4; the rating will be verified by the oral surgeon at time of surgery.

Age between 16-40.

ASA status 1 or 2, deemed in good general health (able to tolerate outpatient conscious sedation safely).

Willing to return at 24 hours for extraction of 1 tooth and be willing to wait up to 6 hours for post op observation following tooth extraction.

Willing to return another 48 hours later for final sensory testing.

EXCLUSION CRITERIA:

ASA status 3-5 and Emergency operation (E) that do not get a physician clearance; i.e. systemic disturbances that limits the patient's activity.

Pregnant or breast-feeding mothers.

Allergy to investigational drugs or to red chili peppers.

Chronically use of analgesics (not limited to, but including: non-steroidal anti-inflammatory medications, steroids, anti-depressants, anti-convulsants).

Presence of chronic disease (e.g. cardiovascular disease, liver disease, kidney disease, diabetes, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 162
Dates: Start 2001-01; Study Completion 2004-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Baranowski R, Lynn B, Pini A. The effects of locally applied capsaicin on conduction in cutaneous nerves in four mammalian species. Br J Pharmacol. 1986 Oct;89(2):267-76. doi: 10.1111/j.1476-5381.1986.tb10256.x. PMID 3779210
- [Background] Berger A, Henderson M, Nadoolman W, Duffy V, Cooper D, Saberski L, Bartoshuk L. Oral capsaicin provides temporary relief for oral mucositis pain secondary to chemotherapy/radiation therapy. J Pain Symptom Manage. 1995 Apr;10(3):243-8. doi: 10.1016/0885-3924(94)00130-D. PMID 7629418
- [Background] Caterina MJ, Schumacher MA, Tominaga M, Rosen TA, Levine JD, Julius D. The capsaicin receptor: a heat-activated ion channel in the pain pathway. Nature. 1997 Oct 23;389(6653):816-24. doi: 10.1038/39807. PMID 9349813